CLINICAL TRIAL: NCT00680875
Title: Intranet-based Tobacco Prevention Program for Children
Acronym: Intranet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CA98555
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Health Promotion; Tobacco Smoking
Keywords: School Based Services; Prevention; Children
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 5th and 6th grade students who attend schools randomly assigned to the intervention condition.
  Interventions: Behavioral: Click City
- Usual Curriculum (No Intervention): 5th and 6th grade students attending schools randomly assigned to the usual curriculum control condition.

INTERVENTIONS:
Behavioral: Click City — School-based intranet delivery of tobacco use prevention program for 5th and 6th graders using interactive and engaging game-like multi-media technology.
  Other Names: Tobacco Free Town
  Arms: Intervention

SUMMARY:
The purpose of this research is to create an effective, disseminable, and exciting computer-based tobacco prevention program for 5th and 6th grade students. The goal of this school-based program is to decrease children's behavioral intentions and willingness to use tobacco, and to prevent or delay their initiation of tobacco use.

We will augment the 5th grade program with a booster program in 6th grade, and evaluate the long-term efficacy of the entire tobacco prevention program by conducting a randomized controlled trial in elementary and middle schools.

DETAILED DESCRIPTION:
The aims of this randomized trail are as follows:

* Conduct a randomized trial to assess the effectiveness of the Tobacco Free Town (TFT) program at preventing or delaying initiation of tobacco by 7th grade, and decreasing behavioral intentions and willingness to use tobacco, as compared to the usual tobacco-prevention curriculum implemented in schools. The TFT program consists of 17 effective components delivered in eight sessions over a four-week period in 5th grade with two booster sessions delivered within a one-week period in 6th grade.
* Develop and test the effectiveness of 7 components to include in the booster sessions in 6th grade using an iterative development process including qualitative evaluation using focus and user groups, and culminating in a quantitative evaluation assessing the effectiveness of individual program components.
* Develop a program guide for teachers to accompany the program and develop parent newsletters for teachers to send home with students after each session.
* Examine change from 5th to 7th grade in the mechanisms that the TFT program is designed to target, and assess if these cognitive mechanisms serve to mediate the effects of the program on smoking outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 5th and 6th grade students attending participating public schools in six counties within a one hour drive of Eugene

Exclusion Criteria:

* Children must be able to read and understand English.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3225 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Self reported cigarette and smokeless tobacco use | 2 years

SECONDARY OUTCOMES:
Intention and willingness to smoke cigarettes or chew smokeless tobacco in the future. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Judy A Andrews, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States